CLINICAL TRIAL: NCT01530620
Title: Efficacy and Tolerability of Propiverine Hydrochloride Extended Release (ER) Compared to Immediate Release (IR) in Patients With Neurogenic Detrusor Overactivity. A Randomized, Double Blind, Parallel Group, Multicenter Clinical Trial
Brief Title: Efficacy and Tolerability of Propiverine Hydrochloride in Patients With Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: APOGEPHA Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8405010
Record Dates: First submitted 2012-02-02; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Neurogenic Urinary Bladder Disorder; Urinary Bladder, Neurogenic; Bladder Disorder, Neurogenic; Urinary Bladder Disorder, Neurogenic; Neurogenic Bladder Disorder; Urinary Bladder Neurogenic Dysfunction; Urologic Diseases; Overactive Detrusor Function; Urinary Incontinence
Keywords: Antimuscarinics; Neurogenic bladder; Propiverine; Urodynamics
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urologic Diseases; Urinary Bladder, Overactive; Urinary Incontinence | interventions — propiverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propiverine hydrochloride ER (Experimental): 45 mg
  Interventions: Drug: Propiverine hydrochloride ER (extended release)
- Propiverine hydrochloride IR (Active Comparator): 15 mg
  Interventions: Drug: Propiverine hydrochloride IR (immediate release)

INTERVENTIONS:
Drug: Propiverine hydrochloride ER (extended release) — 45 mg capsule (1x1/d)
  Other Names: Mictonorm UNO 45; Detrunorm XL 45
  Arms: Propiverine hydrochloride ER
Drug: Propiverine hydrochloride IR (immediate release) — 15 mg tablet (3x1/d)
  Other Names: Mictonorm; Detrunorm
  Arms: Propiverine hydrochloride IR

SUMMARY:
The purpose of this clinical study is to compare efficacy and safety of propiverine hydrochloride extended and immediate release formulations in patients suffering from neurogenic detrusor overactivity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian patients aged ≥18 and ≤70 years
* Voluntarily signed informed consent
* Neurogenic detrusor overactivity with occurrence of reflex detrusor contractions
* Reflex volume of ≤250 mL
* Intact reflex arcs in the area of segments S2-S4

Exclusion Criteria:

* Patients suffering from multiple sclerosis under unstable conditions
* Augmented reflex bladder
* Patients with increased residual urine (≥20 % of the maximum bladder capacity), in whom catheterization is not possible
* Acute urinary tract infection
* Electrostimulation therapy (within 4 weeks propir to Visit 1)
* Anomalies of the lower genitourinary tract (e.g. ectopic ureters, fistulas, urethral stenosis)
* Radiation bladder, interstitial cystitis, bladder calculi, bladder carcinoma
* Surgery of the lower genitourinary tract within the last 6 months (e.g. prostatectomy, hysterectomy, tumor surgery)
* Pre-existing medical contraindications for anticholinergics
* Cardiac insufficiency (NYHA stage III/ IV)
* Therapy with botulinum toxin within the last 12 months
* Evidence of severe renal, hepatic or metabolic disorders
* History of drug or alcohol abuse
* Concomitant medication known to have a potential to interfere with the trial medication
* Known hypersensitivity to Propiverine hydrochloride or excipients contained in the trial medication, respectively
* Pregnant or breast-feeding women, or women of childbearing potential without using any reliable contraceptive method
* Patients with impaired co-operation or who are unable to understand the nature, scope and possible consequences of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-12; Primary Completion 2005-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Reflex volume (cystometry) | three weeks
  Change in reflex volume compared to baseline and compared between the two treatment arms

SECONDARY OUTCOMES:
Leak point pressure | three weeks
  Change in LPP compared to baseline and compared between the two treatment arms
Leak point volume | three weeks
  Change in LPV compared to baseline and compared between the two treatment arms
Maximum detrusor pressure | three weeks
  Change in maximum p det compared to baseline and compared between the two treatment arms
Maximum cystometric capacity | three weeks
  Change in maximum cystometric capacity compared to baseline and compared between the two treatment arms
Bladder compliance | three weeks
  Change in compliance compared to baseline and compared between the two treatment arms
Change in number of incontinence episodes | three weeks
  Change of incontinence episodes compared to baseline and compared between the two treatment arms
State of Well-Being Questionnaire | three weeks
  Change of well-beeing compared to baseline and compared between the two treatment arms
Post void residual volume | three weeks
  Change in PVR compared to baseline and compared between the two treatment arms
Incidence and severity of adverse events | three weeks
  occurrences and intensity of adverse events or withdrawals over the whole treatment period

CONTACTS AND LOCATIONS:
Locations (3):
- Graz, Austria
- Hagenow, Germany
- Bucharest, Romania